CLINICAL TRIAL: NCT03187158
Title: Factors Affecting Early Adult Lung Function
Acronym: FEAL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Sponsor
Other Study IDs: MLP5502
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Early Adult Lung Function; Small Airway Disease; Metabolic Syndrome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Metabolic Syndrome | interventions — Spirometry; Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pune Maternal Nutrition Cohort: Study has been planned on the F1 generation of the mothers recruited under the PMNS study at Diabetes Unit, KEM-Pune. Data on maternal nutrition, exposures and anthropometry have been collected, in the F1 generation. This study will be adding cross sectional lung function measurement, biochemical analyses for nutritional, immunological and inflammatory biomarkers.
  Interventions: Diagnostic Test: Forced Oscillation Technique
- New Delhi Birth Cohort: Study has been planned on the F1 generation of the mothers recruited under the New Delhi Birth Cohort in New Delhi, India. Data on maternal nutrition, exposures and anthropometry have been collected, in the F1 generation, the study will be adding cross sectional lung function measurement, biochemical analyses for nutritional, immunological and inflammatory biomarkers.
  Interventions: Diagnostic Test: Forced Oscillation Technique

INTERVENTIONS:
Diagnostic Test: Forced Oscillation Technique — F.O.T. method can be used to assess obstruction in the large and small peripheral airways , Changes in lung volumes will be measured using a digital spirometer . Every participant will be asked to sit straight, seal the mouthpiece completely with their lips, breathe in fully, blow as hard as possible into the mouthpiece, emptying the lungs completely., Whole blood collected on site (20 mL from every participant, for about 23 metabolites) will be separated into cells and serum. A detailed questionnaire assessing respiratory health, demographic data, habits, and environmental exposure has been developed and validated by Chest Research Foundation.
  Other Names: Spirometry; Questionnaire; Biochemical analysis of nutritional, immunological and inflammatory biomarkers

SUMMARY:
Attainment of peak healthy lung function during the 18-26 yr window is a strong determinant of the rate of lung function decline during the later years of life. The attainment of a healthy peak lung function is mediated by pre and peri natal exposures ( in utero environment and nutrition) and exposure to environmental toxicants and nutrition during childhood and early adulthood. Towards this Indian birth cohorts, having collected comprehensive data on maternal nutrition and anthropometry can provide invaluable insight into the factors affecting lung function growth and their effect sizes in the Indian population. Therefore, in this observational study, the Investigator will be collecting data on lung function, current nutritional and environmental exposures and linking it to pre and peri natal data of the same participants in order to understand lung function growth and the reasons for an early decline in the Indian population, using a life course approach.

DETAILED DESCRIPTION:
Introduction:

Attainment of peak healthy lung function during the 18-26 yr window is a strong determinant of the rate of lung function decline during the later years of life. The attainment of a healthy peak lung function is mediated by pre and peri natal exposures ( in utero environment and nutrition) and exposure to environmental toxicants and nutrition during childhood and early adulthood. Towards this Indian birth cohorts, having collected comprehensive data on maternal nutrition and anthropometry can provide invaluable insight into the factors affecting lung function growth and their effect sizes in the Indian population. Therefore, in this observational study, the Investigator will be collecting data on lung function, current nutritional and environmental exposures and linking it to pre and peri natal data of the same participants in order to understand lung function growth and the reasons for an early decline in the Indian population, using a life course approach.

Sampling:

F1 generation of previously registered Indian Birth Cohorts, having collected comprehensive data on maternal exposures, nutrition and anthropometry.

Techniques Employed:

Spirometry , Forced OscillationTechnique, Anthropometry, Questionnaire, Biochemical analysis of nutritional, immunomodulatory and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* 18-30 years
* Mothers registered in the birth cohort
* Able to perform IOS and Spirometry

Exclusion Criteria:

* Major systemic diseases like cardiac or renal problems
* Clinically significant anemia
* Bone deformity of chest or spine
* muscular weakness
* Otherwise unable to participate in spirometry

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Both birth cohorts,will be instrumental in understanding the link between intergenerational nutrition, early life exposures metabolism and lung health, particularly in rapidly developing lungs. Subjects have already been enrolled in the cohort. Complete datasets of offspring, now aged around 18-30 years, are available through this study, starting from pre-natal environment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test | 12-18 months
  To ascertain whether healthy peak lung function values have been attained
Forced oscillation technique | 12-18 months
  To ascertain the magnitude of airway resistance and study the prevalence of small airway disease

SECONDARY OUTCOMES:
Serum biochemistry | 12-18 months
  To study nutritional, immunological and inflammatory biomarkers correlated with both lung function and metabolic syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Council of Scientific and Industrial Research-Institute of Genomics and Integrative Biology, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Participant data sets and/or documents to be shared : Lung function data, biomarker data, retrospective maternal anthropometry data will be shared as a complete dataset, but with a participant ID which will be delinked from actual participant identity. The ID will only be linked to the participant in the event that an abnormality is detected and the participant may require intervention. Data will be shared via a common excel sheet available to all investigators.